CLINICAL TRIAL: NCT05582330
Title: Turkish Cultural Adaptation, Validation and Reliability Study of Telephone Based ABILOCO-Stroke
Brief Title: Turkish Version of Telephone Based ABILOCO-Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Ünal, Assos. Prof., Pamukkale University
Other Study IDs: 13.10.2022/abiloco
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Cultural Adaptation; Stroke; Reliability; Validity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cultural adaptation, reliability and validity — Cross-cultural Adaptation, Reliability and Validity of the Turkish Version of Telephone Based ABILOCO-Stroke

SUMMARY:
The aims of this study were to perform cultural adaptation of the telephone based ABILOCO-stroke instrument and provide information regarding the factor structure, reliability and validity of the instrument in Turkish speaking patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* hemiparetic individuals who were ≥ 18 years of age
* were at least 4 weeks after the onset of the stroke
* able to walk with or without assistive devices.

Exclusion Criteria:

* cognitive impairments
* aphasia
* any other non-stroke-related conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Telephone Based ABILOCO-Stroke | 10 minutes
  ABILOCO is a measure of locomotion ability for adults with stroke survivors.

IPD SHARING:
Plan to Share IPD: No